CLINICAL TRIAL: NCT01313338
Title: Cognitive Representation, Emotional Responses and Hospitalization Experience in Predicting Decision Making for Receiving Treatment Among Patients With Acute Coronary Syndrome
Brief Title: Experience in Predicting Decision Making for Receiving Treatment in Acute Coronary Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Pimpa Thepphawan, Mahidol university
Other Study IDs: 114/2552(EC3)
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute coronary syndrome

SUMMARY:
The purpose of this study is to examine the predictability of cognitive representation, emotional responses, and hospitalization experience toward the decision to receive treatment of the acute coronary syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute coronary syndrome
* Patients who had first experience or recurrent acute coronary syndrome

Exclusion Criteria:

* Still have chest pain within 24 hours ago
* Cognition or communication disorder or having psychotic or neurologic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome patients
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pimpa Thepphawan, M.Sc, Principal Investigator — Mahidol University
Locations (1):
- Mahidol Univesity, Bangkoknoi, Bangkok, Thailand